CLINICAL TRIAL: NCT00657813
Title: Evaluation of [123I] MNI-330 and Single Photon Emission Computed Tomography (SPECT) as a Marker of Beta-amyloid Protein Deposition in Subjects With Alzheimer Disease in Comparison to Healthy Subjects
Brief Title: Evaluation of [123I] MNI-330 and SPECT as a Marker of Beta-amyloid Protein Deposition
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Data did not evidence [123I]MNI-330 as a useful tool in the detection of AD.
Sponsor: Institute for Neurodegenerative Disorders (Other)
Collaborators: Molecular NeuroImaging (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MNI-330-01
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; SPECT
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Access [123I]MNI-330 and SPECT Imaging (Experimental)
  Interventions: Drug: MNI-330 as a brain SPECT tracer of Beta-Amyloid

INTERVENTIONS:
Drug: MNI-330 as a brain SPECT tracer of Beta-Amyloid — Each subject will receive a bolus injection targeted to be 5 miCi and not to exceed 5.5 mCi of MNI-330. Following injection serial dynamic imaging will be obtained over 8 hrs.

SUMMARY:
The main objectives of this proposal are as follows:

To assess the dynamic uptake and washout of 123-I MNI-330, a potential imaging biomarker for β-amyloid burden in brain, using single photon emission computed tomography (SPECT) in similarly aged Alzheimer's (AD) subjects and healthy controls

To perform blood metabolite characterization of 123-I MNI-330 in healthy and AD subjects to determine the metabolic fate and nature of metabolites in assessment of 123-I MNI-330 as a single photon computed tomography (SPECT) brain imaging agent

Evaluate the test/retest reproducibility of 123-I MNI-330 and SPECT in AD subjects and healthy controls

DETAILED DESCRIPTION:
The underlying goal of this study is to assess 123-I MNI-330 SPECT imaging as a tool to detect ß-amyloid deposition in the brain of AD research participants and age- and gender-matched healthy subjects. All study procedures will be conducted at the Institute for Neurodegenerative Disorders (IND) and Molecular NeuroImaging (MNI) in New Haven, CT. Approximately 10 patients with Alzheimers disease (AD) and 6 healthy controls (within +/- 2 years) will be recruited to participate in this study. Healthy controls will be examined to ensure that there is no evidence of neurodegenerative changes including cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

Alzheimer's Subject Selection. Subjects who have a clinical diagnosis of mild to moderate Alzheimer's disease will be recruited for this study. The following criteria will be met for inclusion of AD subjects in this study:

* The participant is 50 years or older.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of Alzheimer's disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria.
* Mini-Mental Status Exam score < 25.
* Modified Hachinski Ischemia Scale score of ≤ 4.
* Geriatric Depression Scales (GDS) ≤ 10.
* For females, non-child bearing potential or negative urine and blood pregnancy test on day of 123-I MNI-330 injection.

Healthy Control Subject Selection. Healthy control subjects who have no neurological disease will be recruited for this study. The following criteria will be met for inclusion of healthy control subjects in this study:

* The participant is 50 years or older.
* Written informed consent is obtained.
* Negative history of neurological or psychiatric illness based on evaluation by a research physician.
* Mini-Mental Status Exam score ≥28.
* For females, non-child bearing potential or negative urine and blood pregnancy test on day of 123-I MNI-330 injection.

Exclusion Criteria:

Alzheimer's subjects will be excluded from participation for the following reasons:

* The subject has signs or symptoms of another neurodegenerative disease including Parkinson's disease, diffuse Lewy body dementia, or history of significant cerebrovascular disease.
* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Pregnancy

Healthy control subjects will be excluded from participation for the following reasons:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject has any disorder that may interfere with drug absorption distribution, metabolism, or excretion (including gastrointestinal surgery).
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09-30 (Actual); Study Completion 2008-09-30 (Actual)

PRIMARY OUTCOMES:
The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, 123-I MNI-330. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States